CLINICAL TRIAL: NCT02394782
Title: A Prospective, Observational, International, Multi-center Study to Measure the Relationship Between Relapse and Adherence in Relapsing-Remitting Multiple Sclerosis (RRMS) Patients Treated With Rebismart®2.0 + MSdialog™, Assessing Quality of Life (ADHERQOL)
Brief Title: Observational Study of Rebismart®2.0 + MSdialog™ in Subjects With Remitting Multiple Sclerosis (ADHERQOL)
Acronym: ADHERQOL
Status: Terminated | Type: Observational
Why Stopped: lower than anticipated recruitment rate
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200136-591
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: Multiple sclerosis, relapsing-remitting; Rebif; Interferon beta-1a; RebiSmart®2.0; MSdialog™
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Relapsing-remitting Multiple Sclerosis
  Interventions: Device: RebiSmart®2.0; Device: MSdialog™

INTERVENTIONS:
Device: RebiSmart®2.0 — Rebif (interferon beta-1a) will be administered by RebiSmart®2.0 as specified in Summary of Product Characteristics.
Device: MSdialog™ — Rebif (interferon beta-1a) will be administered by MSdialog™ as specified in Summary of Product Characteristics.

SUMMARY:
This is a 24-month, observational, prospective, multinational, multicenter study to determine the relationship between the relapse (percentage of relapse free subjects) and adherence in subjects diagnosed with RRMS treated with Rebif (interferon beta-1a) using the RebiSmart®2.0 and MSdialog™.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RRMS according to McDonald criteria 2010
* Relapse free within 30 days before Baseline data collection
* Treatment with Rebif for 6 months or more prior to informed consent
* Already using RebiSmart®2.0 + MSdialog™ for patient reported outcome (PRO) assessments (at least once prior to informed consent)
* Females of childbearing potential must be willing to use appropriate contraception for the duration of the study
* EDSS score less than (<) 6
* Written informed consent obtained prior to any protocol-required data collection

Exclusion Criteria:

* Participation in other studies within 30 days before Baseline
* Female who is pregnant or breast feeding
* Significant psychiatric symptoms that, in the opinion of the Investigator, would impact subject ability to comply with treatment (as per standard clinical practice)
* Any contraindication for Interferon (IFN) beta-1a therapy as per Summary of Product Characteristics (SPC)
* Administration of any Multiple Sclerosis (MS) therapy, other than Rebif, within 6 months prior to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating sites will identify and recruit eligible subjects using appropriate recruitment strategies in accordance with any local approvals/regulations for observational studies e.g. via clinics, referrals, advertisements, patient databases etc.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Relapse-free Subjects | Up to 24 months
  Relapse is defined as an increase of 2 points in at least one functional system of the expanded disability status scale (EDSS) or an increase of 1 point in at least two functional systems (excluding changes in bowel or bladder function or cognition) in the absence of fever, lasting for at least 24 hours and to have been preceded by at least 30 days of clinical stability or improvement.

SECONDARY OUTCOMES:
Annualized Relapse Rate | Months 12 and 24
  Annualized relapse rate is calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25.
Multiple Sclerosis International Quality of Life (MusiQoL) and Multiple Sclerosis Quality of Life Inventory (MSQLI) Subscale Scores for MSdialog™ | Up to 24 months
  Normalized scores are calculated in the range of 0 - 100; where 0 = the worst QoL status and 100 = the best QoL status (as self-assessed by the subject).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany